CLINICAL TRIAL: NCT01566890
Title: Effect of Adenosine 2A Receptor Agonist Regadenoson on Microvascular Blood Flow in Sickle Cell Anemia
Brief Title: Microvascular Blood Flow in Sickle Cell Anemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Versiti Blood Health (Other)
Collaborators: Medical College of Wisconsin (Other); La Jolla Institute for Allergy & Immunology (Other); University of Illinois at Chicago (Other); Oregon Health and Science University (Other); Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Joshua Field, Principal Investigator, Versiti Blood Health
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: DD2011101
Record Dates: First submitted 2012-03-28; First posted 2012-03-29 (Estimated); Results first posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Sickle Cell Disease; Sickle Cell Anemia
Keywords: sickle cell; sickle cell crisis; sickle cell pain crisis; vaso-occlusive crisis; vaso-occlusion; sickle cell anemia; sickle cell disease; genetic diseases; adenosine 2A Receptor Agonists; Lexiscan; Regadenoson; contrast-enhanced ultrasound; Hydroxyurea
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises; Genetic Diseases, Inborn | interventions — regadenoson

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Regadenoson ARM (Experimental): Adult subjects with sickle cell anemia will receive a regadenoson infusion with contrast-enhanced ultrasound
  Interventions: Drug: regadenoson infusion with contrast-enhanced ultrasound
- Sickle Cell Controls ARM (Other): Adult subjects with sickle cell anemia will receive contrast-enhanced ultrasound
  Interventions: Procedure: contrast-enhanced ultrasound
- Sickle Cell CEU ARM (Other): Adults subjects with sickle cell anemia will receive contrast-enhanced ultrasound
  Interventions: Procedure: contrast-enhanced ultrasound
- Healthy Control ARM (Other): Healthy African American control subjects without sickle cell anemia will receive contrast-enhanced ultrasound
  Interventions: Procedure: contrast-enhanced ultrasound
- Technique Optimization Controls (Other): Healthy volunteers will undergo contrast-enhanced ultrasound.
  Interventions: Procedure: contrast-enhanced ultrasound

INTERVENTIONS:
Drug: regadenoson infusion with contrast-enhanced ultrasound — Subjects who are not having a pain crisis receive a 24-hour infusion of regadenoson. Contrast-enhanced ultrasound will be performed four times during the 24 hour regadenoson infusion
  Other Names: Lexiscan; regadenoson
  Arms: Regadenoson ARM
Procedure: contrast-enhanced ultrasound — Subjects who are not having a pain crisis will have contrast-enhanced ultrasound performed up to four times over a two-day period. Time points will resemble the time course used for the Regadenoson Arm, although no investigational drug will be given.
  Arms: Sickle Cell Controls ARM
Procedure: contrast-enhanced ultrasound — Contrast-enhanced ultrasound will be performed on adults with sickle cell anemia at baseline who are not having a pain crisis and performed again during a pain crisis
  Arms: Sickle Cell CEU ARM
Procedure: contrast-enhanced ultrasound — Contrast-enhanced ultrasound will be performed on healthy control subjects at baseline, on the first day of the study and 30 days later
  Arms: Healthy Control ARM
Procedure: contrast-enhanced ultrasound — Contrast-enhanced ultrasound will be performed on healthy volunteers (Technique Optimization Controls)
  Arms: Technique Optimization Controls

SUMMARY:
Sickle cell disease (SCD) is an inherited blood disorder that causes the red blood cells to change their shape from a round shape to a half-moon/crescent or sickled shape. Sickle-shaped cells can cause problems by getting stuck in blood vessels, blocking blood flow, and can cause inflammation and injury to important body parts. There are no specific treatments that improve this condition and promote blood flow hindered by sickle cell blockages. Another big challenge in managing sickle cell disease is that there are no good measures to determine changes and improvements in blood flow.

Contrast-enhanced ultrasound is a technique currently used to detect blood flow in the heart, muscles, and other organs. It is extremely sensitive and can detect blood flow in the smallest of blood vessels. It would be very useful in helping healthcare providers know whether treatment strategies are improving blood flow during sickle cell blockages.

The hypothesis is that contrast-enhanced ultrasound will be a feasible tool for determining changes in blood flow of subjects with sickle cell disease.

DETAILED DESCRIPTION:
Sickle cell disease is an inherited blood disorder that affects one of every 400 African-Americans newborns in the United States. Sickle cell disease causes the red blood cells to change their shape from a round shape to a half-moon sickle shape. Individuals who have sickle cell disease have a different type of protein that carries oxygen in the blood (hemoglobin) than individuals without sickle cell disease. This different type of hemoglobin makes the red blood cell change into a crescent shape under certain conditions. Sickle shaped cells are a problem because the often get stuck on blood vessels blocking the flow of blood, and cause inflammation and injury to important areas of the body. These symptoms can lead to a painful occurrence called a "sickle cell crisis". Many individuals have to be admitted into the hospital because of the pain caused by a sickle cell crisis.

Regadenoson is a drug that may help prevent inflammation and injury caused by the sickle shaped cells. This drug is approved by the FDA to be used as a bolus during a heart stress test in people unable to exercise enough to put stress on the heart by making it beat faster. In a recent Phase I study, a safe dose for regadenoson was determined for adults with sickle cell disease. This dose was given by a slow IV infusion for a 24-48 hour period.

Hydroxyurea is the only FDA approved drug for the treatment of sickle cell disease. Hydroxyurea is a pill taken orally and works well but is not useful during a severe sickle cell crisis.

In this study researchers will use a new method, contrast-enhanced ultrasound (CEU), to visualize tiny blood vessels in cardiac and skeletal muscle. Changes in CEU measurements before, during and after administration of regadenoson will be examined. Contrast-enhanced ultrasounds will also be performed in individuals who are not having a sickle cell crisis. Some of those individuals will also undergo CEU while they are having a sickle cell crisis to compare those measurements . Lastly CEU results will be compared between individuals with sickle cell anemia and healthy African-Americans. These CEU's will be used to determine if there are changes in the blood flow of tiny blood vessels in certain conditions.

This study wants to know if this new method of contrast-enhanced ultrasound will be a useful tool for physicians to use in individuals with sickle cell anemia. The researchers also want to determine if this new method of CEU can be used to reveal if some treatments for sickle cell anemia work better than others.

ELIGIBILITY:
Inclusion Criteria:

Regadenoson ARM Inclusion Criteria:

* Diagnosis of sickle cell anemia confirmed by hemoglobin analysis
* Ages 18 to 70 years
* Subjects must have laboratory indices as outlined by the protocol
* Reliable IV access as determined by physician

Sickle Cell Controls ARM Inclusion Criteria:

* Diagnosis of sickle cell anemia confirmed by hemoglobin analysis
* Ages 18 to 70 years

Sickle Cell CEU ARM Inclusion Criteria:

* Diagnosis of sickle cell anemia, confirmed by hemoglobin analysis
* Males and females age 18-70 years

Healthy Control ARM Inclusion Criteria:

* African American
* Ages 18 to 70 years

Technique Optimization Control ARM Inclusion Criteria:

-Ages 18 to 70 years

Exclusion Criteria:

Regadenoson ARM Exclusion Criteria

* Hospitalization, emergency department visit or self-reported crisis within last 2 weeks for any reason or 4 weeks from acute chest syndrome
* Current physician diagnosis of active asthma (within last 12 months) or current use of asthma medications
* Second or third degree AV block or sinus node dysfunction
* Known or suspected right to left sided cardiac shunts
* History of a bleeding diathesis
* History of clinically overt stroke
* History of severe hypertension not adequately controlled with anti-hypertensive medications
* Receiving chronic anti-coagulation or anti-platelet therapy
* History of metastatic cancer
* Receiving other investigational study agents, or have received a study agent in the last 30 days
* Uncontrolled intercurrent illness
* Pregnant or breastfeeding women
* Subjects who have a HIV infection
* Subjects who have had a hematopoietic stem cell transplant
* Subjects who are taking medications that may interact with the investigational agent
* Prior hypersensitivity reactions to either regadenoson or ultrasound contrast agents

Sickle Cell Controls Exclusion Criteria:

* Hospitalization, emergency department visit or self-reported crisis within last 2 weeks for any reason or 4 weeks from acute chest syndrome
* Known pregnancy
* Known history of HIV
* Known or suspected right to left sided cardiac shunts
* Receiving other investigational study agents, or have received a study agent within the last 30 days
* Subjects who have had a hematopoietic stem cell transplant
* Prior hypersensitivity reactions to ultrasound contrast agents
* History of severe hypertension not adequately controlled with anti-hypertensive medications
* Uncontrolled intercurrent illness

Sickle Cell CEU ARM Exclusion Criteria:

* Pregnant women
* Subjects who have a HIV infection
* History of stem cell transplant
* Current involvement in a therapeutic clinical trial
* Known or suspected right to left sided cardiac shunts
* Prior hypersensitivity reactions to ultrasound contrast agents
* History of severe hypertension not adequately controlled with anti-hypertensive medications
* Uncontrolled intercurrent illness

Healthy Control ARM Exclusion Criteria:

* Sickle cell disease or sickle cell trait
* Known or suspected right to left sided cardiac shunts
* Diagnosis of type 1 or type 2 diabetes mellitus
* Hypertension
* History or current diagnosis of dyslipidemia or taking lipid lowering drugs
* Diagnosis of coronary artery disease or peripheral vascular disease
* Body weight greater than 10% of ideal weight
* Uncontrolled intercurrent illness
* Pregnant or breastfeeding women
* Subjects who have a HIV infection
* Prior hypersensitivity reactions to ultrasound contrast agents

Technique Optimization Control ARM Exclusion Criteria:

* Known sickle cell disease or sickle cell trait
* Known or suspected right to left sided cardiac shunts
* Uncontrolled intercurrent illness
* Known pregnant or breastfeeding women
* Prior hypersensitivity reactions to ultrasound contrast agents

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2012-07; Primary Completion 2019-07-05 (Actual); Study Completion 2020-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua J Field, MD, MS, Principal Investigator — Medical College of Wisconsin; Jonathon Lindner, MD, Principal Investigator — Oregon Health and Sciences University
Locations (2):
- United States (2):
  - The University of Illinois, Chicago, Illinois
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Background] Ashley-Koch A, Yang Q, Olney RS. Sickle hemoglobin (HbS) allele and sickle cell disease: a HuGE review. Am J Epidemiol. 2000 May 1;151(9):839-45. doi: 10.1093/oxfordjournals.aje.a010288. PMID 10791557
- [Background] Charache S, Terrin ML, Moore RD, Dover GJ, Barton FB, Eckert SV, McMahon RP, Bonds DR. Effect of hydroxyurea on the frequency of painful crises in sickle cell anemia. Investigators of the Multicenter Study of Hydroxyurea in Sickle Cell Anemia. N Engl J Med. 1995 May 18;332(20):1317-22. doi: 10.1056/NEJM199505183322001. PMID 7715639
- [Background] {Field, 2011 #10443}Field, J. J., D. G. Nathan, et al. (2011).
- [Derived] Belcik JT, Davidson BP, Xie A, Wu MD, Yadava M, Qi Y, Liang S, Chon CR, Ammi AY, Field J, Harmann L, Chilian WM, Linden J, Lindner JR. Augmentation of Muscle Blood Flow by Ultrasound Cavitation Is Mediated by ATP and Purinergic Signaling. Circulation. 2017 Mar 28;135(13):1240-1252. doi: 10.1161/CIRCULATIONAHA.116.024826. Epub 2017 Feb 7. PMID 28174191

RESULTS

PARTICIPANT FLOW:
Groups:
- Sickle Cell Crisis ARM: Adult subjects who had a sickle cell crisis
  Adults subjects with sickle cell anemia will receive contrast-enhanced ultrasound
  contrast-enhanced ultrasound: Contrast-enhanced ultrasound will be performed on adults with sickle cell anemia at baseline who are not having a pain crisis and performed again during a pain crisis
- Healthy Controls: Healthy African American control subjects without sickle cell anemia will receive contrast-enhanced ultrasound
Period: Overall Study
Arm/Group | Regadenoson ARM | Sickle Cell Controls ARM | Sickle Cell Crisis ARM | Healthy Controls | Technique Optimization Controls
Started | 32 | 10 | 21 | 21 | 7
Completed | 21 | 6 | 10 | 7 | 0
Not Completed | 11 | 4 | 11 | 14 | 7
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 1 | 1 | 0
Not completed — Screen failure | 6 | 0 | 1 | 1 | 0
Not completed — Incomplete CEU data | 1 | 3 | 5 | 8 | 0
Not completed — Lost to Follow-up | 0 | 0 | 4 | 4 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 7

BASELINE CHARACTERISTICS:
Population: For this study, baseline measures of heart rate and blood pressure were taken 5-10 minutes apart, prior to drug administration and/or (in control groups) a contrast enhanced ultrasound was performed. Baseline was defined as the subject doing well, reporting no more than baseline pain, and being at least 2 weeks from a hospitalization or emergency department visit. Healthy Controls and Technique Optimization Controls are not listed as these groups were intended to determine intravariability.
Groups:
- Healthy Controls: Healthy African American control subjects without sickle cell anemia will receive contrast-enhanced ultrasound.
  They were not included in the analysis due to the number of participants who did not complete the study (therefore no meaningful ultrasounds to interpret).
- Technique Optimization Controls: Healthy volunteers will undergo contrast-enhanced ultrasound.
  There was no data collected for this arm.
- Total: Total of all reporting groups
Arm/Group | Regadenoson ARM | Sickle Cell Controls ARM | Sickle Cell Crisis ARM | Healthy Controls | Technique Optimization Controls | Total
Number analyzed (Participants) | 20 | 6 | 6 | 7 | 0 | 39
Age, Continuous [Median (Full Range); unit: years] | 25 [20 to 46] | 35 [27 to 48] | 26 [22 to 40] | 26 [20 to 46] |  | 26 [20 to 48]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 7 |  | 7
  Male | 20 | 6 | 6 | 0 |  | 32
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20 | 6 | 6 | 7 |  | 39

OUTCOME MEASURES:

1. Primary Outcome: Microvascular Blood Flow Rate Change
Description: Primary outcome measure will be a 40% increase in skeletal muscle microvascular blood flow when 24 hour measurements are compared to baseline in subjects receiving Regadenoson. We took measurements in patients who received Regadenoson, as well as Sickle Cell controls. Both arms had microvascular blood flow (volume x velocity) measured at baseline and 24-hours, and those values were compared. A change ratio of >1 means that the flow rate increased at 24 hours and a change ratio of <1 means that the flow rate decreased at 24 hours.
Time Frame: Between baseline and 24 hours
Population: There were 20 participants in the Regadenoson arm, and 6 participants acted as sickle cell controls. Sickle Cell Crisis ARM is not included because arm was not measured by CEUS in a similar timeframe as Regadenoson ARM and Sickle Cell Controls ARM, as indicated in Results Baseline Characteristics Arm/Group Description for Sickle Cell Crisis ARM.
Measure: Median (Full Range); unit: Ratio of change
Arm/Group | Regadenoson ARM | Sickle Cell Controls ARM
Number analyzed (Participants) | 20 | 6
Ratio of change | 1.09 [0.39 to 4.12] | 0.86 [0.24 to 2.82]

2. Secondary Outcome: MVBF Ratio of Change During a Pain Crisis
Description: We planned to examine differences in microvascular blood flow using contrast-enhanced ultrasound (CEU) in adults with sickle cell anemia age 18 and older at baseline state compared to a pain crisis. We were measuring changes in microvascular blood flow in subjects with sickle cell anemia during a pain crisis by examining differences in microvascular blood flow using contrast-enhanced ultrasound at a baseline state, and comparing those measurements to contrast-enhanced ultrasound measurements during a pain crisis. A change ratio of >1 means that the flow rate increased during a pain crisis and a change ratio of <1 means that the flow rate decreased during a pain crisis.
Time Frame: Between baseline and between 7-30 days after pain crisis, if feasible
Measure: Median (Full Range); unit: Ratio of change
Groups:
- Sickle Cell Crisis ARM: Adult subjects who had a sickle cell crisis
  Contrast-enhanced ultrasound will be performed on adults with sickle cell anemia at baseline who are not having a pain crisis and performed again during a pain crisis
Arm/Group | Sickle Cell Crisis ARM
Number analyzed (Participants) | 6
Ratio of change | 0.65 [0.60 to 0.95]

3. Secondary Outcome: Microvascular Blood Flow in Sickle Cell Anemia Subjects Versus Control Subjects
Description: Examine microvascular blood flow using contrast-enhanced ultrasounds in adult subjects with sickle cell anemia compared to microvascular blood flow of healthy African-American adults
Time Frame: 5 years
Population: African American controls subjects were enrolled. The ultrasounds were not able to be examined and therefore no data generated to provide.
Arm/Group | Healthy Controls
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from the time participants signed consent until they completed their last study visit (about 30 days).
Description: The definition of an adverse event did not differ from the clinicaltrials.gov definition.
Arm/Group | Regadenoson ARM | Sickle Cell Controls ARM | Sickle Cell CEU ARM | Healthy Control ARM | Technique Optimization Controls
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/10 | 0/21 | 0/21 | 0/7
Serious Adverse Events (participants affected / at risk) | 5/32 | 0/10 | 3/21 | 0/21 | 0/7
Other Adverse Events (participants affected / at risk) | 16/32 | 3/10 | 4/21 | 1/21 | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regadenoson ARM (N=32) | Sickle Cell Controls ARM (N=10) | Sickle Cell CEU ARM (N=21) | Healthy Control ARM (N=21) | Technique Optimization Controls (N=7)
Vaso Occlusive Crisis (Vascular disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Vaso-Occlusive Crisis consistent with Sickle Cell Pain Crisis
Severe Pain (Vascular disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) — Severe Diffuse or Targeted Pain that begins after CEU Procedure consistent with description in package insert
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regadenoson ARM (N=32) | Sickle Cell Controls ARM (N=10) | Sickle Cell CEU ARM (N=21) | Healthy Control ARM (N=21) | Technique Optimization Controls (N=7)
Pain (General disorders) | 13 (17) | 1 (1) | 3 (3) | 0 (0) | 0 (0) — Pain
Nausea and/or Vomiting (Gastrointestinal disorders) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — joint stifness
Cheilitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysguesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Blurred Vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot flash (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
As with any study, ours had limitations. The most significant limitation was our small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-02): https://cdn.clinicaltrials.gov/large-docs/90/NCT01566890/Prot_SAP_000.pdf